CLINICAL TRIAL: NCT04998669
Title: Phase 2, Single-arm, Open-label, Study of Loncastuximab Tesirine in Combination With Rituximab in Patients With Relapsed or Refractory Follicular Lymphoma
Brief Title: Loncastuximab Tesirine in Combination With Rituximab in Patients With Relapsed or Refractory Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Juan P. Alderuccio, MD (Other)
Collaborators: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor-Investigator, Juan P. Alderuccio, MD, Associate Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20201130
Record Dates: First submitted 2021-08-07; First posted 2021-08-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — loncastuximab tesirine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Loncastuximab tesirine + Rituximab (Experimental): During the 12-week Induction Phase (Cycles 1 to 4), participants will receive loncastuximab tesirine on days 1 of each 3-week cycle for Cycles 1 through 4; and rituximab on days 1, 8, 15 of Cycle 1 and day 1 of Cycle 2.
  Maintenance Phase 1 (Cycle 5) is 8 weeks: Participants achieving complete response (CR) or partial response (PR) during the Induction Phase will receive loncastuximab tesirine once every 3-weeks; and rituximab once during week 7 or 8. Participants achieving a response of Stable Disease (SD) or Progressive Disease (PD) will be taken off treatment.
  Maintenance Phase 2 (Cycles 6 and 7) is 16 weeks:
  * Participants achieving CR during Maintenance Phase 1 receive rituximab once during week 7 or 8 of Cycles 6 and 7.
  * Participants achieving PR during Maintenance Phase 1 receive loncastuximab tesirine once every 3-weeks over each 8 week cycle; and rituximab once during week 7 or 8 of Cycles 6 and 7.
  * Participants achieving SD or PD will be taken off treatment.
  Interventions: Drug: Loncastuximab tesirine; Drug: Rituximab

INTERVENTIONS:
Drug: Loncastuximab tesirine — Induction Phase (Cycles 1 through 4):
  * 150 μg/Kg of loncastuximab tesirine administered via intravenous infusion (given as per treatment guidelines) on Days 1 of a 3-week cycle during Cycles 1 and 2.
  * 75 μg/Kg of loncastuximab tesirine administered via intravenous infusion (given as per treatment guidelines) on Days 1 of a 3-week cycle during Cycles 3 and 4.
  Maintenance Phase 1 (Cycle 5): For participants achieving CR or PR, 75 μg/Kg of loncastuximab tesirine administered via intravenous infusion (given as per treatment guidelines). on Day 1 on Week 1, 4, 7 of a 8-week cycle.
  Maintenance Phase 2 (Cycle 6 & 7): For participants achieving PR, 75 μg/Kg of loncastuximab tesirine administered via intravenous infusion (given as per treatment guidelines) on Day 1 on Week 1, 4, 7 of a 8-week cycle.
  Other Names: ADCT-402
Drug: Rituximab — Induction Phase (Cycles 1 through 4): 375 mg/m2 rituximab on days 1, 8, 15 of cycle 1 and day 1 of cycle 2 via intravenous infusion (given as per treatment guidelines) or subcutaneous 1400 mg/23,400 units hyaluronidase during Cycles 1 and 2, per discretion of treating physician. Rituximab will not be administered during Cycles 3 and 4.
  Maintenance Phase 1 (Cycle 5): Participants achieving a response of PR or CR will receive 375 mg/m2 rituximab during week 1 of a 8-week cycle via intravenous infusion (given as per treatment guidelines) or subcutaneous 1400 mg/23,400 units hyaluronidase, per discretion of treating physician.
  Maintenance Phase 2 (Cycles 6 and 7): Participants achieving a response of PR or CR will receive 375 mg/m2 rituximab during week 1 of each 8-week cycle via intravenous infusion (given as per treatment guidelines) or subcutaneous 1400 mg/23,400 units hyaluronidase, per discretion of treating physician.
  Other Names: Rituxan

SUMMARY:
The purpose of this research is to see if Loncastuximab Tesirine in combination with Rituximab will result in higher complete response rate when given to treat follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Patients must have histologic confirmation of Follicular Lymphoma (FL) (grade 1, 2 and 3A). Note: Participants who have received previous CD19-directed therapy must have a biopsy which shows CD19 expression after completion of the CD19-directed therapy.
3. Patients with relapsed or refractory FL previously treated with ≥1 line of systemic therapy having ≥ 1 Groupe d'Etude des Lymphomes (GELF) criteria for therapy, or Progression of Diseases within 24 months (POD24), or second relapse.
4. Baseline FDG-PET/CT scans must demonstrate positive lesions compatible with CT defined anatomical tumor sites. Patients should have at least one measurable site of disease per Lugano classification.
5. Patient should have ≥ 1 Groupe d'Etude des Lymphomes (GELF) criteria for treatment initiation).

   * Involvement of ≥3 nodal sites, each with diameter of ≥3 cm
   * Any nodal or extranodal tumor mass with a diameter of ≥7 cm
   * B symptoms (fever ≥ 38 degrees Celsius of unclear etiology, night sweats, weight loss > 10% within the prior 6 months).
   * Risk of local compressive symptoms that may result in organ compromise
   * Splenomegaly or splenic lesion without splenomegaly
   * Leukopenia (leukocytes < 1000/mm3)
   * Leukemia (> 5.000 lymphoma cells/mm3)
   * Bone lesions detected on FDG-PET/CT; or
6. Progression or relapse within 24 months of frontline treatment in patients previously treated with ≥1 line of systemic therapy; or
7. Second FL relapse/progression after ≥1 line of systemic therapy. These patients will be eligible independently of GELF criteria and POD24.
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
9. Life expectancy of greater than 6 weeks.
10. Patients must have normal organ and marrow function as defined below,

    * Absolute neutrophil count ≥1000/mm3 (unless due to lymphoma involvement of the bone marrow or spleen).
    * Platelets ≥100,000/mm3 or ≥ 60,000/mm3 in case of bone marrow involvement by lymphoma.
    * Hemoglobin ≥ 10 g/dL or ≥8 g/dL in case of bone marrow involvement by lymphoma.
    * Total bilirubin < 1.5 x within normal institutional limits (unless due to lymphoma involvement of liver or a known history of Gilbert's disease).
    * Gamma-Glutamyl Transpeptidase (GGT)/Aspartate Aminotransferase (AST)/(SGOT)/Alanine Aminotransferase (ALT)(SGPT) ≤ 2.5 × institutional upper limit of normal.
    * Creatinine within normal institutional limits, or creatinine clearance ≥30 ml/min/1.7m^2 for patients with creatinine levels above institutional normal (unless due to lymphoma).

Exclusion Criteria:

1. FL grade 3B or transformed FL.
2. [Removed]
3. ≥ 6 lines of systemic immunochemotherapy for treatment of FL.
4. Patients with clinically significant pleural effusions and/or ascites requiring drainage or associated with shortness of breath.
5. Patients receiving any other investigational agents.
6. Patients with known central nervous system involvement of lymphoma.
7. Uncontrolled intercurrent illness such as: history of Myocardial Infarction (MI) in the last 6 months, congestive heart failure New York Heart Association (NYHA) Class III-IV, uncontrolled or symptomatic arrhythmia, stroke in last 6 months, liver cirrhosis, and autoimmune disorder requiring immunosuppression or long-term corticosteroids (>10 mg daily prednisone equivalent).
8. Breastfeeding or pregnant women.
9. Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody will need a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.) Hepatitis C antibody positive patients are eligible if PCR is negative. Hepatitis B core antibody (+) patients without evidence of HBsAg or Hep B PCR (+) are eligible with appropriate Hepatitis B reactivation prophylaxis.
10. History of Human immunodeficiency virus (HIV) infection. Note: HIV screening test is optional
11. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving Complete Response (CR) | 12 weeks
  Complete Response rate will be reported as the number of participants achieving complete response (CR) to study therapy. Response to therapy will be assessed using Fluorodeoxyglucose (FDG)-Positron Emission Tomography (PET) (FDG-PET)/ Computerized Tomography (CT) following Lugano 2014 criteria by week 12 of treatment.

SECONDARY OUTCOMES:
Number of participants achieving CR or PR | Week 12
  Overall response rate (ORR) will be reported as the number of participants achieving complete response (CR) or partial response (PR) by the end of the induction phase, week 12. Response to therapy will be assessed using Fluorodeoxyglucose (FDG)-Positron Emission Tomography (PET) (FDG-PET)/ Computerized Tomography (CT) following Lugano 2014 criteria.
Incidence of Treatment-Related Adverse Events | Up to 13 months
  Safety of the intervention will be reported as the incidence of treatment-related toxicity, including serious adverse events (SAEs) and adverse events (AEs), in study participants using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.
Progression-free Survival (PFS) | Up to 3 years
  Progression-Free Survival (PFS) is defined as the elapsed time from the date of starting treatment (Cycle 1 Day 1) until disease progression or death (whichever occur first).
Overall Survival (OS) | Up to 3 years
  Overall survival (OS) will be defined as the elapsed time from the date of starting treatment (Cycle 1 Day 1) until death.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Alderuccio, MD, Principal Investigator — University of Miami
Locations (5):
- United States (5):
  - Florida Cancer Specialists and Research Institute, Fort Myers, Florida
  - University of Miami, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Allegheny Health Network, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alderuccio JP, Alencar AJ, Schatz JH, Kuker RA, Pongas G, Reis IM, Lekakis LJ, Spiegel JY, Sandoval-Sus J, Beitinjaneh A, Stanchina MD, Trabolsi A, Lossos IS, Rosenblatt JD, Lessen DS, Moskowitz CH. Loncastuximab tesirine with rituximab in patients with relapsed or refractory follicular lymphoma: a single-centre, single-arm, phase 2 trial. Lancet Haematol. 2025 Jan;12(1):e23-e34. doi: 10.1016/S2352-3026(24)00345-4. Epub 2024 Dec 7. PMID 39662486